CLINICAL TRIAL: NCT00393783
Title: Xenogeneic HER2/Neu DNA Immunization for Patients With Metastatic and High Risk Breast Cancer: A Phase I Study to Assess Safety and Immunogenicity
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-101
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic; HER2; 04-101
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Trastuzumab

ARMS (1):
- 1 (Experimental): HER2 ECD DNA.
  Interventions: Biological: MAB HER 2 (HERCEPTIN)

INTERVENTIONS:
Biological: MAB HER 2 (HERCEPTIN) — Rat HER2 DNA will be delivered intramuscularly at four different dose levels (0.5mg, 1mg, 3mg, or 6mg) during weeks 1, 4, 7, 10 and 13 for five injections.

SUMMARY:
The purpose of this study is to evaluate whether the injection of HER2/neu DNA is safe and stimulates an immune response.

The immune system consists of different kinds of cells and substances which help fight against infections and inflammation in the body. These antibodies and T-cells are part of the immune system that may also help to fight against tumor cells. One way to make antibodies and stimulate T-cells is to inject the patient with a preparation which contains material that may stimulate the immune system. This process is called an immunization. We are trying to immunize the patient against HER2/neu. In order to participate in this trial, the tumor must have a large amount of HER2/neu on its surface. The injection that the patient will receive in this trial is a piece of DNA made in bacteria which contains the gene for rat HER2. DNA is material which contains the information needed to produce many substances in the body. The HER2 gene encodes for a protein known as HER2.

ELIGIBILITY:
Breast cancer patients with AJCC Stage III or metastatic (AJCC Stage IV) disease that over-express HER2 will potentially be eligible for this trial. Patients may have measurable disease, evaluable disease or be without evidence of disease. They may be receiving hormonal therapy and they may have already received trastuzumab (Herceptin) or be receiving trastuzumab during this study.

Inclusion Criteria:

Patients must have ALL of the features listed below:

* AJCC Stage IV breast cancer (histologically confirmed) with no evidence of disease or stable disease. Patients may be either off therapy or on hormone therapy and/or trastuzumab.

OR AJCC Stage III breast cancer < or = to 36 months post completion of adjuvant therapy.

* Pathology slides must be reviewed by the Department of Pathology at MSKCC.
* HER2 over-expression by FISH or by staining 3+ on immunohistochemistry in either the primary or metastatic tumor.
* Karnofsky performance status > or = to 80%.
* Patients must have recovered from the toxicity of any prior therapy, and not received major surgery, radiation therapy, or chemotherapy for at least 4 weeks prior to entry into the trial. (Ongoing hormonal therapy and/or trastuzumab administration is permitted.)
* Age > 18 years

Exclusion Criteria:

* Pregnancy (Women of child bearing potential must not be pregnant and have a normal pregnancy test within 2 weeks of starting treatment.) Woman who may yet bear children and sexually active men must be using appropriate contraception during the course of this study. Patients must be counseled not to become pregnant during the study. Patients must also be counseled that injection of HER2 may have unknown affects on the viability of a future fetus.
* Nursing
* Prior cumulative doxorubicin dose > 360 mg/m2
* Prior cumulative epirubicin dose > 600 mg/m2
* Other active cancers (within the prior five years, excluding non-melanoma skin cancer).
* Inadequate organ function as defined by any of the following:

  * total white blood cell count of < 3,000 cells/mm3
  * platelet count < 100,000/mm3
  * serum creatinine > 1.5 x upper limit of normal
  * aspartate aminotransferase (AST) > 2 x the upper limit of normal
* History of cardiac disease as defined by any of the following:

  * any prior myocardial infarction
  * history of documented congestive heart failure
  * left ventricular ejection fraction below the normal institutional range
  * use of medications for treatment of angina pectoris
  * any prior arrhythmia or cardiac valvular disease requiring medication or clinically significant
* History of known immunodeficiency or autoimmune disease.
* Any use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to respond immunologically to vaccines is grounds for exclusion, at the discretion of the Principal Investigator or co-Principal Investigators.
* Previous breast cancer vaccine exposure
* Active CNS or leptomeningeal tumor
* Active infection requiring antibiotic treatment
* Anticipated survival of less than 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose over four dose levels | 13 weeks

SECONDARY OUTCOMES:
A secondary endpoint is to observe patients for any evidence of anti-tumor effect. | at week 19 or at the discretion of the physician

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org